CLINICAL TRIAL: NCT06614192
Title: AndroMETa-CRC-064: An Open Label, Randomized, Controlled, Global Phase 3 Study Comparing Telisotuzumab Adizutecan (ABBV-400) Monotherapy to LONSURF (Trifluridine and Tipiracil) Plus Bevacizumab in Subjects With Refractory Metastatic Colorectal Cancer Expressing c-Met Protein Level Above a Defined Cutoff
Brief Title: A Study Assessing Adverse Events and Disease Activity When Comparing Intravenously (IV) Infused ABBV-400 to Trifluridine and Tipiracil (LONSURF) Oral Tablets Plus IV Infused Bevacizumab in Adult Participants With c-Met Protein Above Cutoff Level Above Refractory Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-064; 2024-512804-20-00 (Other: EU CT)
Record Dates: First submitted 2024-09-25; First posted 2024-09-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Telisotuzumab Adizutecan; ABBV-400; Trifluridine; Tipiracil; LONSURF; Bevacizumab; AndroMETa-CRC-064
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1: Telisotuzumab Adizutecan Dose A (Experimental): Participants will receive telisotuzumab adizutecan dose A, as part of the approximately 4 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Stage 1: Telisotuzumab Adizutecan Dose B (Experimental): Participants will receive telisotuzumab adizutecan dose B, as part of the approximately 4 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Stage 2: Telisotuzumab Adizutecan Optimal Dose (Experimental): Participants will receive the optimal dose of telisotuzumab adizutecan, as part of the approximately 4 year study duration.
  Interventions: Drug: Telisotuzumab Adizutecan
- Stage 2: Standard of Care (SOC) (Experimental): Participants will receive the SOC, as part of the approximately 4 year study duration.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Arms: Stage 1: Telisotuzumab Adizutecan Dose A; Stage 1: Telisotuzumab Adizutecan Dose B; Stage 2: Telisotuzumab Adizutecan Optimal Dose
Drug: Trifluridine/Tipiracil — Oral Tablet
  Other Names: LONSURF
  Arms: Stage 2: Standard of Care (SOC)
Drug: Bevacizumab — IV Infusion
  Arms: Stage 2: Standard of Care (SOC)

SUMMARY:
Colorectal cancer (CRC) is the third most common type of cancer diagnosed worldwide and in China. The purpose of this study is to assess adverse events disease activity when comparing intravenously (IV) infused telisotuzumab adizutecan to trifluridine and tipiracil (LONSURF) oral tablets plus IV infused bevacizumab in adult participants with c-Met protein above cutoff level refractory metastatic colorectal cancer (mCRC).

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of CRC. Participants are put into treatment arms as part of 2 stages. Each treatment arm in stage 1 receives a different dose of telisotuzumab adizutecan. Each treatment arm in stage 2 receives the optimal dose of telisotuzumab adizutecan or LONSURF plus bevacizumab. Up to approximately 460 adult participants with c-Met protein above cutoff level refractory mCRC, will be enrolled in the study in approximately 160 sites in 15-20 countries.

In stage 1, participants will receive intravenously (IV) infused telisotuzumab adizutecan dose A or B. In stage 2, participants will receive the optimal dose of IV infused telisotuzumab adizutecan or the standard of care (SOC), LONSURF oral tablets plus IV infused bevacizumab. The total study duration will be approximately 4 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >= 12 weeks per investigator assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 during the screening period prior to the first dose of the study drug.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

Exclusion Criteria:

* Prior systemic regimen containing c-MET targeting antibody/bispecific or Antibody Drug Conjugate (c-Met targeting Antibody Drug Conjugate [ADC]).
* History of allergic reactions or hypersensitivity to bevacizumab or any of its excipients, or to compounds similar to trifluridine/tipiracil.
* Active infection as noted in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Percentage of Participants with Adverse Events (AE)s | Up to a Maximum of 4 Years
  An AE is defined as any untoward medical occurrence, inappropriate patient management decision, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, users or other persons whether or not related to the investigational drug.
Stage 1: Percentage of Participants with Clinically Significant Vital Sign Measurements as Assessed by the Investigator | Up to a Maximum of 4 Years
  Vital signs are defined as determinations of systolic and diastolic blood pressure, pulse rate, respiratory rate, oxygen saturation (SpO2), and body temperature will be obtained at visits.
Stage 1: Percentage of Participants with Clinically Significant Electrocardiograms (ECGs) Findings as Assessed by the Investigator | Up to a Maximum of 4 Years
  Percentage of participants with clinically significant ECGs findings as assessed by the investigator.
Stage 1: Percentage of Participants with Clinically Significant Laboratory Values (Chemistry, Hematology, Coagulation, and Urinalysis) as Assessed by the Investigator | Up to a Maximum of 4 Years
  Percentage of participants with clinically significant laboratory values (hematology, chemistry, coagulation, and urinalysis) as assessed by the investigator.
Stage 1 and Stage 2: Objective Response (OR) as Assessed by Blinded Independent Central Review (BICR) | Up to a Maximum of 4 Years
  OR is defined as confirmed complete response (CR) or confirmed partial response (PR) as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
Stage 2: Overall Survival (OS) | Up to a Maximum of 4 Years
  OS is defined as the time from randomization to the event of death from any cause.

SECONDARY OUTCOMES:
Stage 1 and Stage 2: Progression Free Survival (PFS) as Assessed by BICR | Up to a Maximum of 4 Years
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by BICR or death from any cause, whichever occurs earlier.
Stage 1: OS | Up to a Maximum of 4 Years
  OS is defined as the time from randomization to the event of death from any cause
Stage 1 and Stage 2: Duration of Response (DOR) as Assessed by BICR | Up to a Maximum of 4 Years
  DOR is defined as the time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST v1.1 as determined by BICR or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
Stage 1 and Stage 2: Disease Control (DC) as Assessed by BICR | Up to a Maximum of 4 Years
  DC is defined as best overall response of confirmed CR or confirmed PR, or stable disease (SD) based on RECIST, version 1.1 as determined by BICR.
Stage 1 and Stage 2: OR as Assessed by Investigator | Up to a Maximum of 4 Years
  OR is defined as confirmed CR or confirmed PR as assessed by investigator per RECIST, version 1.1.
Stage 1 and Stage 2: PFS as Assessed by Investigator | Up to a Maximum of 4 Years
  PFS is defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 as determined by investigator or death from any cause, whichever occurs earlier.
Stage 1 and Stage 2: DOR as Assessed by Investigator | Up to a Maximum of 4 Years
  DOR is defined as the time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST v1.1 as determined by BICR or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
Stage 1: Maximum Observed Serum (or Plasma, for Payload) Concentration (Cmax) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Maximum observed serum (or plasma, for payload) concentration for telisotuzumab adizutecan.
Stage 1: Time to Cmax (Tmax) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Time to Cmax for telisotuzumab adizutecan.
Stage 1: Terminal Elimination Half-Life (t1/2) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Terminal elimination half-life for telisotuzumab adizutecan.
Stage 1: Area Under the Serum (or Plasma, for Payload) Concentration Versus Time Curve (AUC) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Area under the serum (or plasma, for payload) concentration versus time curve will be determined using noncompartmental methods for total antibody for telisotuzumab adizutecan.
Stage 1: Antibody Drug Conjugate (ADC) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Antibody drug conjugate for telisotuzumab adizutecan.
Stage 1: Unconjugated Topoisomerase 1 (Top1) Inhibitor Payload for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Unconjugated Top1 inhibitor payload for telisotuzumab adizutecan.
Stage 1: Incidence of Anti-Drug Antibodies (ADAs) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Incidence of anti-drug antibodies for telisotuzumab adizutecan.
Stage 1: Neutralizing Anti-Drug Antibodies (nADAs) for Telisotuzumab Adizutecan | Up to a Maximum of 4 Years
  Neutralizing anti-drug antibodies for telisotuzumab adizutecan.
Stage 2: Change from Baseline at C5D1 in Physical Functioning as Measured by the Physical Functioning Domain of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/Quality of Life (QoL) scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Stage 2: Change from Baseline at C7D1 (Standard of Care [SOC] Arm) in Physical Functioning as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Stage 2: Change from Baseline at C5D1 in in Diarrhea as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/Quality of Life (QoL) scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Stage 2: Change from Baseline at C7D1 (SOC Arm) in Diarrhea as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Stage 2: Change from Baseline at C5D1 in in Global Health Status (GHS)/QoL as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/Quality of Life (QoL) scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).
Stage 2: Change from Baseline at C7D1 (SOC Arm) in GHS/QoL as Measured by the Physical Functioning Domain of the EORTC QLQ-C30 | Up to a Maximum of 4 Years
  The EORTC QLQ-C30 is a 30-item patient-reported questionnaire composed of both multi-item and single scales including 5 functional scales (physical, role, emotional, social, and cognitive), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale ranging from 1 to 4 (1 = Not at All, 2 = A Little, 3 = Quite a Bit, and 4 = Very Much).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (51):
- United States (24):
  - City of Hope National Medical Center /ID# 267875, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 270655, Irvine, California
  - USC Norris Comprehensive Cancer Center /ID# 268131, Los Angeles, California
  - Lutheran Medical Center- Cancer Centers of Colorado /ID# 268175, Golden, Colorado
  - Yale New Haven Hospital /ID# 269125, New Haven, Connecticut
  - AdventHealth Orlando /ID# 267970, Orlando, Florida
  - Winship Cancer Institute of Emory University /ID# 266884, Atlanta, Georgia
  - St. Luke's Cancer Institute: Boise /ID# 268095, Boise, Idaho
  - Northwestern Memorial Hospital /ID# 268610, Chicago, Illinois
  - Hope And Healing Cancer Services /ID# 268541, Hinsdale, Illinois
  - Springfield Clinic - First /ID# 268666, Springfield, Illinois
  - Community Cancer Center North /ID# 267965, Indianapolis, Indiana
  - Hattiesburg Clinic /ID# 267860, Hattiesburg, Mississippi
  - Washington University /ID# 267872, St Louis, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana /ID# 268185, Billings, Montana
  - Rutgers Cancer Institute of New Jersey /ID# 268056, New Brunswick, New Jersey
  - University of North Carolina Medical Center /ID# 266879, Chapel Hill, North Carolina
  - Duke University Medical Center /ID# 267966, Durham, North Carolina
  - Avera Cancer Institute - Sioux Falls /ID# 268074, Sioux Falls, South Dakota
  - West Cancer Center and Research Institute - Germantown /ID# 268619, Germantown, Tennessee
  - University of Texas - Southwestern Medical Center /ID# 268241, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center /ID# 268098, Houston, Texas
  - Millennium Research & Clinical Development /ID# 268400, Houston, Texas
  - University of Virginia /ID# 268108, Charlottesville, Virginia
- Mater Hospital Brisbane /ID# 268360, South Brisbane, Queensland, Australia
- Israel (6):
  - The Chaim Sheba Medical Center /ID# 267741, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 267578, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 267739, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 267579, Jerusalem
  - Rabin Medical Center /ID# 267740, Petah Tikva
  - Assuta Medical Center /ID# 267745, Tel Aviv
- Japan (5):
  - Aichi Cancer Center /ID# 268237, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 268236, Kashiwa-shi, Chiba
  - The University of Osaka Hospital /ID# 268743, Suita-shi, Osaka
  - Saitama Prefectural Cancer Center /ID# 268706, Kitaadachi-gun, Saitama
  - National Cancer Center Hospital /ID# 268713, Chuo-Ku, Tokyo
- Pan American Center for Oncology Trials /ID# 267888, Rio Piedras, Puerto Rico
- South Korea (5):
  - Seoul National University Bundang Hospital /ID# 268592, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 268719, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 268718, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 268717, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 268720, Seoul, Seoul Teugbyeolsi
- Taiwan (9):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 267638, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 267627, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 270464, Changhua City, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 267635, Kaohsiung City
  - China Medical University Hospital /ID# 267631, Taichung
  - Taichung Veterans General Hospital /ID# 270467, Taichung
  - National Cheng Kung University Hospital /ID# 270468, Tainan
  - Taipei Veterans General Hospital /ID# 267628, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 267637, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-064